CLINICAL TRIAL: NCT04279327
Title: Diagnostic Value of Cell Block Immunohistochemistry in Effusion Cytology
Brief Title: Cell Block Immunohistochemistry in Effusion Cytology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliaa Elhosainy Mohammad Mahmoud, Associate Lecturer, Assiut University
Other Study IDs: immuno-cytology001
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Effusion Pleural; Ascites; Pericardial Effusion
Keywords: immunohistochemistry; cytology; moc 31 monoclonal antibody, human
MeSH Terms: conditions — Pleural Effusion; Ascites; Pericardial Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: cytology positive for malignancy
- controls: cytology negative for malignancy

SUMMARY:
Cytology is usually the first step in investigating serous effusions, to either detect or exclude an underlying malignancy. This study will try to answer the need for improved diagnostic yield of cytologic examination by cell block technique and immunohistochemical testing of three markers which are EZH2, Claudin-4 and MOC-31.

DETAILED DESCRIPTION:
This is a prospective study that will be conducted at the pathology lab of Assiut University Hospital. The study will include effusion specimens (pleural, peritoneal & pericardial) and the aspirated fluid will be examined for physical characters e.g. color and appearance.

The sample will be divided into 2 equal parts: one for conventional smear preparation, and the other for cell block. A minimum of 2 thin smears will be prepared and stained with Papanicolou stain.

Cell block sections of 4-6 μ thickness will be prepared and stained with the hematoxylin and eosin stain (H&E).

For immunohistochemistry, cell blocks will be used. Expression of claudin 4, EZH2, and MOC-31 will be evaluated in benign and malignant cells by using immunoperoxidase technique.

ELIGIBILITY:
Inclusion Criteria:

* all cases with serous effusion of unknown aetiology including ascites, pleural or pericardial effusions.

Exclusion Criteria:

* No exclusion criteria from the histopathologist perspective, i.e. all cases that undergone diagnostic aspiration are eligible for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all cases that have serous effusion of undiagnosed underlying aetiology.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of EZH2 | within 48 hours
  sensitivity and specificity of EZH2 for diagnosis of malignancy
Diagnostic performance of claudin4 | within 48 hours
  sensitivity and specificity of claudin-4 for diagnosis of malignancy
Diagnostic performance of MOC-31 | within 48 hours
  sensitivity and specificity of MOC-31 for diagnosis of malignancy

SECONDARY OUTCOMES:
Prevalence of malignancy among cases presenting with effusion | one year
  percentage of cases diagnosed with malignancy among all cases presenting with effusion

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa EM Mahmoud, MSc, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sundling KE, Cibas ES. Ancillary studies in pleural, pericardial, and peritoneal effusion cytology. Cancer Cytopathol. 2018 Aug;126 Suppl 8:590-598. doi: 10.1002/cncy.22021. PMID 30156768